CLINICAL TRIAL: NCT07352163
Title: Effects of Training With Proprioceptive Neuromuscular Facilitation on Vertical Jump Performance and Postural Stability in Male Basketball Players
Brief Title: PNF Training Effects on Jump and Balance in Basketball Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Keskin (Other)
Responsible Party: Sponsor-Investigator, Merve Keskin, Research Assistant, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0762
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Physical Performance and Postural Stability in Healthy Male Basketball Players
Keywords: Proprioceptive Neuromuscular Facilitation Postural Balance, Athletic Performance, Basketball, Male
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation (Active Comparator): Participants will be included in a 6-week program in which they will perform lower extremity proprioceptive neuromuscular facilitation patterns 3 days a week for a total of approximately 20-30 minutes.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation
- Control Group (No Intervention): No intervention will be performed on the control group.

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — During training, rhythmic initiation and combined isotonic PNF techniques will be applied. Rhythmic initiation will be performed through passive, active-assisted, and resistive phases to facilitate motor learning and coordination, with each phase repeated three times (one set). Combined isotonic exercises aim to enhance muscle activation and neuromuscular control by sequentially applying concentric, isometric, and eccentric contractions within a single continuous movement. Moderate manual resistance will be provided by the therapist at the beginning, middle, and end of the range of motion. Combined isotonic exercises will be performed bilaterally for 6-10 repetitions and 3-4 sets, with 60 seconds of rest between sets, in accordance with participant tolerance.
  Arms: Proprioceptive Neuromuscular Facilitation

SUMMARY:
The purpose of this study is to examine the effect of PNF applications on vertical jump performance and postural control in male basketball players.

The hypotheses of this study are:

H1: PNF applications affect vertical jump performance in male basketball players.

H2: PNF applications have an effect on postural control in male basketball players.

H3: There is no difference between the PNF group and the control group in terms of the effect of PNF applications on vertical jump performance and postural control in male basketball players.

Participants will be included in a 6-week program based on the group they are assigned to in the randomization. Those in the exercise group will perform lower extremity PNF patterns 3 days a week for a total of approximately 20-30 minutes. No intervention will be performed on the control group. Participants' vertical jump performance and postural control will be assessed twice: before and after the intervention.

DETAILED DESCRIPTION:
This study is planned as a randomized controlled trial. After obtaining ethical committee approval, the study will be conducted on male basketball players within one year. The population of the study consists of male basketball players. The sample of the study will consist of male professional basketball players aged 18-35 who volunteer to participate in the study. To calculate the sample size of the study, a study (14) using similar methods was considered, and based on the hypothesis that the difference between the two groups would have a medium effect size, a two-way variance analysis was performed using the G*Power Version 3.1.9.2 (Franz Faul, Universitat Kiel, Germany) program. The results indicate an effect size of f=0.41, replication = 2, number of groups = 2, correlation between repeated measures = 0.5, Type I error = 0.05, and statistical power = 0.99. This resulted in a sample size of at least 15 patients per group, totaling 30 patients. Participants will be divided into two groups using the block randomization method: the PNF group and the control group. Block randomization will be performed via https://www.sealedenvelope.com/simple-randomiser/v1/lists.

All participants' demographic information will be collected via a form. Participants will be included in a 6-week program based on the group they are assigned to in the randomization. If they are in the exercise group, they will perform lower extremity PNF patterns 3 days a week for a total of approximately 20-30 minutes. Rhythmic initiation and combined isotonic PNF techniques will be used during training. Two basic PNF techniques will be applied during the training process. Rhythmic initiation is performed by gradually and repeatedly performing the movement pattern using passive, active-assisted, and resistive movement phases to improve movement learning and coordination. Each phase of the movement pattern (passive, active-assisted, resistive) will be performed 3 times, for a total of 1 set. The goal of combined isotonic exercises is to increase muscle activation and improve neuromuscular control throughout the targeted lower extremity movement pattern. During the application, sequential manual resistance is applied at different stages of the movement, and all concentric, isometric, and eccentric contractions are performed in a single fluid movement. Resistance is applied in a controlled manner by the therapist at the beginning, middle, and end of the range of motion. Combined isotonic exercises will be performed with 6-10 repetitions and 3-4 sets, with 60 seconds of rest between sets, by sequentially and fluidly applying concentric-isometric-eccentric contractions under moderate manual resistance throughout the target pattern. All techniques will be applied bilaterally in a controlled, standardized manner appropriate to participant tolerance. No intervention will be applied to the control group. Participants' vertical jump performance and postural control will be assessed twice: before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-35,
2. Licensed basketball players,
3. Individuals willing to participate in the study will be included.

Exclusion Criteria:

1. Individuals who have undergone any trauma/surgical procedure within the last 6 months,
2. Individuals with any injury or health condition that could affect the results of the relevant assessments,
3. Individuals with severe-to-moderate local and/or general musculoskeletal pain will not be included.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
VERTICAL JUMP PERFORMANCE | At baseline and from enrollment to the end of treatment at week 6.
  In the vertical jump test, the difference between the height reached while standing and the height reached while jumping (m) will be taken, and anaerobic power data will be calculated from the Lewis Nomogram together with body weight (kilograms).
POSTURAL CONTROL | At baseline and from enrollment to the end of treatment at week 6.
  Postural control assessment will be performed statically and dynamically using the Biodex Balance System SD (Biodex Medical Systems, Inc., Shirley, NY).

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Çiğli, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No